CLINICAL TRIAL: NCT01239849
Title: A Multicenter, Eight Weeks Treatment, Single Step Titration, Open Label Study Assessing the Percentage of Korean Diabetic Dyslipidemic Patients Achieving LDL Cholesterol Target With Atorvastatin Starting Dose 10mg, 20mg, 40mg
Brief Title: Korean AMADEUS Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Bucheon St Mary Hospital, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKimlipid
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2009-02

CONDITIONS: Diabetes Mellitus, Hypercholessterolemia
Keywords: Diabetes Mellitus, Hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus; Hypercholesterolemia | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Atorvastatin, 10mg, 20mg, 40mg — If initial LDL cholesterol between 100~ 129mg/dl then starting dose of Atorvastatin is 10mg, 130~159 mg/dl is 20 mg, 160~220mg/dl is 40mg.
  After 4weeks treatment, if LDL cholesterol is below 100mg/dl then continue starting dose and if not reach below 100mg/dl then titration double dose.
  After 4 weeks treatment, recheck the LDL cholesterol

SUMMARY:
Because Diabetes Mellitus is one of the major risk factors for CV disease and lots of related evidences have been published including CARDS study that showed definite benefit of statin treatment in DM patients and influenced ADA guideline. & NCEP ATP III update. However, there are large unmet medical needs for DM patients who don't reach their target LDL-C level defined NCEPT ATP III update because of physicians usually start with the lowest dose of statin and then titrate to the goal. Thus, we are curious about changing our prescription pattern into more tailored way; selecting starting dose based on the individual risk factors and concomitant status will impact the goal achieving rate for DM patients. Besides that, we are going to find out preliminary data about other markers change; small dense LDL and adiponectine;. Small dense LDL-C is more inflammatory and atherogenic LDL-C that may explain the impact of triglyceride. Adiponectin is another good marker related with obesity and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Korean Diabetes Patients
2. Is ≥ 18 and ≤ 80 years olds
3. Has diagnosis of dyslipidemia
4. Has 100 mg/dl ≤ LDL cholesterol ≤ 220 mg/dl
5. Has triglyceride level ≤ 600 mg/dl
6. Has HbA1c ≤ 12%
7. If female, is postmenopausal, surgically sterilized, or using a reliable methods of birth control considered suitable by the investigator
8. Can discontinue all current antilipidemic medication for the 4 week washout period
9. Has provided written informed consent prior to the initiation of any study procedure

Exclusion Criteria:

1. Is pregnant or lactating
2. Abuse alcohol and/or any other drug
3. Uncontrolled diabetes ( HbA1c > 12% )
4. Has impaired hepatic function, as shown by but not limited to alanine aminotransferase (ALT,SGOT) or aspartate aminotransferase (AST, SGOT) ≥ 2times the upper limit of normal at baseline.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-12 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects in the total LDL cholesterol group achieving their LDL cholesterol target after 8 weeks of treatment. | 8 weeks

SECONDARY OUTCOMES:
1. Percentage of subjects in the total LDL cholesterol group achieving their LDL cholesterol target after 4 weeks of treatment. | 8 weeks
2. Change and percent change from baseline to 4 and 8 weeks of treatment for LDL cholesterol, HDL cholesterol, non-HDL cholesterol, LDL cholesterol/HDL cholesterol ratio, Total cholesterol, Triglyceride subjects in the total group. | 8 weeks
3. Percentage of subjects who achieved LDL cholesterol target with no titration of atorvastatin and after one step titration of atorvastatin | 8 weeks
4. Change and percent change from baseline to 4 and 8 weeks of treatment for small dense LDL cholesterol, adiponectin, hs-CRP | 8 weeks
5. Safety of atorvastatin through laboratory assessment, physical examination, vital signs, and adverse events. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SUNG RAE KIM, A. Professor, Principal Investigator — Bucheon St. Mary Hospital, The Catholic University of Korea
Locations (1):
- Sung Rae Kim, Bucheon-si, Kyeongki, South Korea

REFERENCES:
- [Derived] Son JW, Kim DJ, Lee CB, Oh S, Song KH, Jung CH, Mok JO, Kim JH, Moon MK, Choi KM, Cho JH, Choi SH, Kim SK, Park KS, Kim HS, Kim IJ, Kim YI, Kim HJ, Kim SY, Kim S. Effects of patient-tailored atorvastatin therapy on ameliorating the levels of atherogenic lipids and inflammation beyond lowering low-density lipoprotein cholesterol in patients with type 2 diabetes. J Diabetes Investig. 2013 Sep 13;4(5):466-74. doi: 10.1111/jdi.12074. Epub 2013 Mar 26. PMID 24843697